CLINICAL TRIAL: NCT01232166
Title: Endotracheal Tube Insertion Depth Better Detects Endobronchial Intubation Than Bilateral Auscultation or Observation of Chest Movements - a Prospective Randomised Trial
Brief Title: Which is the Best Bedside Test to Detect Endobronchial Intubation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Univ. Prof. Chiari, Medical University; Department for Anesthesia and General Intensive Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MUW464/2003
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-10

CONDITIONS: Endobronchial Intubation
MeSH Terms: interventions — Auditory Perception; Off-Road Motor Vehicles

STUDY DESIGN:
Who Masked: Investigator

ARMS (8):
- Endobronchial Intubation, Auscultation (Experimental): In this arm, the endotracheal tube will be positioned in the right main stem bronchus under direct visualization through a fiberoptic bronchoscope. The study anesthesiologists will then perform bilateral auscultation of the lungs only, with the patient's thorax and head covered with blankets to blind participants to thorax movements and ETT insertion depth (Group Auscultation, n=20)
  Interventions: Other: Auscultation
- Endobronchial Intubation, Observation (Active Comparator): In this arm, the endotracheal tube (ETT) will be positioned in the right main stem bronchus under direct visualization through a fiberoptic bronchoscope. To determine the position of the ETT the study anesthesiologists will then perform observation and palpation of symmetric chest movements without auscultation of the lungs, with the patient's head covered with blankets to blind participants to ETT insertion depth (Group Observation, n=20);
  Interventions: Other: Observation of symmetric chest movements
- Endobronchial intubation, tube depth (Active Comparator): In this arm, the endotracheal tube (ETT) will be positioned in the right main stem bronchus under direct visualization through a fiberoptic bronchoscope. To determine the position of the ETT the study anesthesiologists will then estimate ETT position by observing the ETT cm scale without lung auscultation, with the patient's thorax covered by blankets to blind participants to thorax movements (Group Tube Depth, n=20)
  Interventions: Other: Tube depth
- Endobronchial intubation, all three (Active Comparator): In this arm, the endotracheal tube (ETT) will be positioned in the right main stem bronchus under direct visualization through a fiberoptic bronchoscope. To determine the position of the ETT the study anesthesiologists will then perform a combination of auscultation, observation and tube depth
  Interventions: Other: All three
- Endotracheal Intubation, Auscultation (Experimental): In this arm, the endotracheal tube will be positioned in the trachea, 2,5-4cm above the carina under direct visualization through a fiberoptic bronchoscope. The study anesthesiologists will then perform bilateral auscultation of the lungs only, with the patient's thorax and head covered with blankets to blind participants to thorax movements and ETT insertion depth (Group Auscultation, n=20)
  Interventions: Other: Auscultation
- Endotracheal Intubation, observation (Active Comparator): In this arm, the endotracheal tube (ETT) will be positioned in the trachea, 2,5-3cm above the carina under direct visualization through a fiberoptic bronchoscope. To determine the position of the ETT the study anesthesiologists will then perform observation and palpation of symmetric chest movements without auscultation of the lungs, with the patient's head covered with blankets to blind participants to ETT insertion depth (Group Observation, n=20);
  Interventions: Other: Observation of symmetric chest movements
- Endotracheal intubation, tube depth (Active Comparator): In this arm, the endotracheal tube (ETT) will be positioned in the trachea, 2,5 - 4 cm above the carina under direct visualization through a fiberoptic bronchoscope. To determine the position of the ETT the study anesthesiologists will then estimate ETT position by observing the ETT cm scale without lung auscultation, with the patient's thorax covered by blankets to blind participants to thorax movements (Group Tube Depth, n=20)
  Interventions: Other: Tube depth
- Endotracheal intubation, all three (Active Comparator): In this arm, the endotracheal tube (ETT) will be positioned 2,5-4cm above the carina under direct visualization through a fiberoptic bronchoscope. To determine the position of the ETT the study anesthesiologists will then perform a combination of auscultation, observation and tube depth
  Interventions: Other: All three

INTERVENTIONS:
Other: Auscultation
  Arms: Endobronchial Intubation, Auscultation; Endotracheal Intubation, Auscultation
Other: Observation of symmetric chest movements
  Arms: Endobronchial Intubation, Observation; Endotracheal Intubation, observation
Other: Tube depth
  Arms: Endobronchial intubation, tube depth; Endotracheal intubation, tube depth
Other: All three
  Arms: Endobronchial intubation, all three; Endotracheal intubation, all three

SUMMARY:
Background: Endotracheal intubation has become a well established standard in protecting the airway during surgical procedures, and in emergency situations. Serious complications can occur from the incorrect placement of an endotracheal tube in a mainstem bronchus. If unrecognized it can lead to hypoxemia secondary to atelectasis of the unventilated lung and hyperinflation of the intubated lung, which can result in barotrauma. As bedside method the golden standard to verify the correct endotracheal tube placement is bilateral ausculation of the chest. However this is not always satisfactory, as breath sounds can be transmitted to the opposite side of the chest in spite of endobronchial intubation. Therefore other clinical tests to verify the correct endotracheal tube placement have become part of daily clinical practice, like observation of symmetric chest movements, and use of the cm markings printed on the endotracheal tube. However so far no study investigated which of these bedside clinical methods works best in detecting an inadvertently placed endobronchial tube in adults. We therefore designed a study to compare three different bedside methods to verify endotracheal or endobronchial tube placement.

Objective: To determine which of four commonly used bedside methods of detecting inadvertent endobronchial intubation in adults has the highest sensitivity and specificity.

Design: Prospective randomized, blinded study. Setting: Tertiary, academic hospital, department of anaesthesia. Participants: 160 consecutive ASA I or II patients, aged 19-75 years, scheduled for elective gynaecological or urological surgery.

Interventions: Patients were randomly assigned to eight study groups. In four groups, an endotracheal tube (ETT) was fiberoptically positioned 2.5-4.0 cm above the carina, whereas in the other four groups the tube was positioned in the right mainstem bronchus. The four groups differed in the bedside test used to verify the position of the endotracheal tube. First-year residents and experienced anaesthesiologists independently performed one of the following randomly assigned bedside tests in each patient in an effort to determine whether the tube was properly positioned in the trachea: 1) bilateral auscultation of the chest (Auscultation); 2) observation and palpation of symmetric chest movements (Observation); 3) estimating the position of the ETT by the insertion depth (Tube Depth); and, 4) a combination of all three mentioned tests (All Three).

Main outcome measures: Correct and incorrect judgements of endotracheal tube (ETT) position as independently assessed by first-year anaesthesia residents and experienced anaesthesiologists with each of the four bedside tests.

ELIGIBILITY:
Inclusion Criteria:

ASA I or II patients, aged 19-75 years, scheduled for elective gynaecological or urological surgery that needs endotracheal intubation.

Exclusion Criteria:

* Pre-existing lung disease, pleural effusion, anticipated difficult airway, known endobronchial or tracheal lesions, or patients at risk for aspiration of gastric contents.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-03; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity/Specificity to detect endobronchial intubation | 1-5 minutes after intubation
  First-year residents and experienced anaesthesiologists independently performe one of four randomly assigned bedside tests in each patient to determine whether the tube was positioned in the trachea or endobronchially

REFERENCES:
- [Derived] Sitzwohl C, Langheinrich A, Schober A, Krafft P, Sessler DI, Herkner H, Gonano C, Weinstabl C, Kettner SC. Endobronchial intubation detected by insertion depth of endotracheal tube, bilateral auscultation, or observation of chest movements: randomised trial. BMJ. 2010 Nov 9;341:c5943. doi: 10.1136/bmj.c5943. PMID 21062875